CLINICAL TRIAL: NCT05165368
Title: Effect of Gluten-Free Dietary Education and Intraneural Facilitation® Therapy on Quality of Life in People With Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5210345
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Neuropathy, Distal Symmetric Polyneuropathy (Manifestation)
Keywords: Intraneural Facilitation® Therapy, Dietary Education, Gluten-free diet, Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Using the block randomization method, patients will be randomly assigned to the INF® Therapy only group or the INF® Therapy+ group. Ten participants will be recruited at a time with 5 randomly assigned to each group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcomes assessor will be blinded to interventional group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraneural Facilitation® Therapy (INF® Therapy) + Dietary Education (Experimental): The INF® Therapy+ group will receive dietary education with weekly follow-up by a physical therapist either in person, or via email or text message. The INF® Therapy+ group will additionally receive meal preparation ideas and sample menus promoting a gluten-free diet.
  Interventions: Other: Intraneural Facilitation® Therapy (INF® Therapy)
- Intraneural Facilitation® Therapy (INF® Therapy) (Active Comparator): INF® Therapy is a manual therapy technique that consists of three components. The first is the pressurization or facilitation hold which biases circulation more consistently in the nerves, which is thought to "pressurize the entire system" The secondary hold attempts to stretch the innervated structure, pulling apart the tough dividing membrane and allowing the pressurized blood flow to transport from the outside "holding" chamber to the endoneurium and push open the closed capillary beds next to the nerve axons. Once capillaries surrounding the nerves are pressurized, the circulation needs to be induced up the neural connective tissue. A separate set of pressure points or "holds" are performed distal to the secondary holds to ensure the circulation is drawn up the inflamed capillary beds using the Bernoulli principle.
  Interventions: Other: INF® Therapy

INTERVENTIONS:
Other: Intraneural Facilitation® Therapy (INF® Therapy) — INF® Therapy plus dietary education with weekly follow-up by a physical therapist. Includes meal preparation ideas and sample menus promoting a gluten-free diet.
  Other Names: INF® Therapy plus Dietary Education
  Arms: Intraneural Facilitation® Therapy (INF® Therapy) + Dietary Education
Other: INF® Therapy — INF® Therapy only (INF® Therapy is a manual therapy technique that consists of three components. The first is the pressurization or facilitation hold which biases circulation more consistently in the nerves, which is thought to "pressurize the entire system" The secondary hold attempts to stretch the innervated structure, pulling apart the tough dividing membrane and allowing the pressurized blood flow to transport from the outside "holding" chamber to the endoneurium and push open the closed capillary beds next to the nerve axons. Once capillaries surrounding the nerves are pressurized, the circulation needs to be induced up the neural connective tissue. A separate set of pressure points or "holds" are performed distal to the secondary holds to ensure the circulation is drawn up the inflamed capillary beds using the Bernoulli principle.)
  Arms: Intraneural Facilitation® Therapy (INF® Therapy)

SUMMARY:
The purpose of this research is to compare the effectiveness of providing dietary education to complement Intraneural Facilitation® Therapy (INF® Therapy) (a physical therapy technique being evaluated that may help improve circulation) versus INF® Therapy only in adults with a type of neuropathy called distal symmetric polyneuropathy (DSPN).

DETAILED DESCRIPTION:
[All participants] First assessment session for research purposes only: Participants will complete the informed consent, VAS pain scale, HIPAA, and medical screening documents. Using the block randomization method, patients will be randomly assigned to the INF® Therapy only group or the INF® Therapy+ group by a research coordinator who will not be conducting any participant assessments. Ten participants will be recruited at a time with five randomly assigned to each of the two groups. Then all participants will be given brief explanations before administration of the questionnaires.

Participants will first be instructed to complete the visual analog scale (VAS) for pain, a subjective measure of pain intensity consisting of a 10-centimeter (cm) line with anchor statements on the left (no pain) and extreme pain on the right. Pain scores will be determined by measuring the distance in cm from "no pain" to the participant's anchor point. Participants who rate their pain level on the visual analog scale (VAS) as greater than seven out of ten level will be excluded from study participation due to poorly controlled pain.

Next, participants will complete a series of self-report questionnaires beginning with the CDAT questionnaire which gathers selected information on frequency of purposeful gluten consumption and self-efficacy to maintain compliance with a gluten-free diet.

The medical screening questionnaire will assess for important comorbid conditions that may influence outcomes.

Next, the PSQI is a clinical questionnaire assessing quality of sleep and sleep disturbances over the past month. The 19-item questionnaire provides seven component scores assessing subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medications, and daytime dysfunction.

Further, the IPAQ-S measures intensity of physical activity and sitting time to estimate total physical activity per week. Computation of the total score for the short form requires summation of the duration (in minutes) and frequency (days) of walking, moderate-intensity and vigorous-intensity activities.

Finally, participants will complete the STAI-form Y which is a definitive clinical measure of state and trait anxiety in adults. Form Y has 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.

All participants will be familiarized to the Neuropad® test and MiniBESTest prior to taking measurements. The Neuropad® test measures sweat production as an indicator for peripheral neuropathy severity in people with type 2 diabetes. The time for the cobalt (II) chloride indicator to complete color change from blue to pink is correlated to severity of nerve conduction impairment: 892±179 seconds in severe nerve conduction impairment, and 1983±386 in those with moderate nerve conduction impairment (P =.01). Sudometrics image analysis software will be utilized to analyze Neuropad® time to color change since it produces continuous outputs to quantify neuropathic severity. The test will be applied between the first and second metatarsal bases, avoiding calloused areas after a standard 10-minute prior period without socks or shoes sitting in a room at a constant 20-25 degrees Celsius. After 10 minutes of test applied, the Neuropad® square will be removed and immediately scanned on a flatbed scanner to capture the color change result. The image will be analyzed using Sudometrics software which produces objective continuous outputs to quantify neuropathic severity.

Next, participants will perform mini balance evaluation system test (Mini-BESTest) which contains 14 tasks under 4 balance-related subcategories of anticipatory (3 items), reactive postural control (3 items), sensory orientation (3 items), and dynamic gait (5 items), and takes approximately 15 minutes to administer. Each item is scored from 0 (unable) to 2 (normal) with a maximum score of 28.

All participants will receive the standard of care INF® Therapy evaluations and treatments for ten sessions total, two sessions per week (visits two through eleven). During the initial INF® Therapy evaluation (visit two), three questionnaires will be administered (Background Information, PQAS, and LENS), and selected data collected for analysis as specified below. An INF® Therapy treatment will follow the INF® Therapy evaluation.

During INF® Therapy treatment sessions (visits three through ten), either a physical therapist or physical therapist assistant will provide INF® Therapy treatments. No research data will be collected during the INF® Therapy treatment sessions.

During the INF® Therapy re-evaluation on visit eleven, the LENS and PQAS questionnaires will be administered as a post assessment.

[To be completed at initial INF® Therapy evaluation only, visit two] Participants will complete the Background Information form (self-report) and the following data will be collected from the form for research purposes as these factors may influence participant outcomes: participant's gender, smoking, peripheral arterial disease (PAD), hypertension (HTN), hypercholesteremia, and consumption of the following medications: statins, gabapentin, or Neurontin.

[To be completed at INF® Therapy initial & re-evaluation, visits two and eleven] The Lower Extremity Neuropathy Scale (LENS) is a combined assessment including patient report of sensory and balance disturbances, and clinician-administered, objective assessment of ankle dorsiflexion strength, vibration and light touch sensitivity, gait mechanics, and balance during conditions of both static single leg stance and dynamic heel-to-toe pattern during gait. Use of the LENS is for INF® Therapy PT evaluation only as part of the standard of care. A separate study for the validation of this tool is in progress. No data from this tool will be collected for the proposed study.

[To be completed at INF® Therapy initial & re-evaluation, visits two and eleven] The Pain Quality Assessment Scale (PQAS) is an adjusted version of the validated Neuropathic Pain Scale and includes 20 pain qualities and descriptors. The tool is validated for detecting changes in pre-post treatment pain quality and spatial characteristics of pain. Four of the 10 new items showed statistically significant (P .0025) pretreatment to post-treatment changes, while nine of the items showed at least a moderate effect size (d > .50).12 The validation study for the original Neuropathic Pain Scale found Pearson correlation coefficients ranging from .04 to .73.13 The majority of these (39 or 87%) were less than 0.50, indicating minimal overlap (i.e., less than 25% of variance) between most items.13 The means and standard deviations between items for patients with diabetic neuropathy ranged from 1.76 to 6.54 (2.27 to 3.75) with excellent significance (p < .01).13

[For INF® Therapy+ group only: The clinical therapists will receive training to standardize the gluten-free dietary (GFD) education to be provided to study participants:

1. Dr. Bussell will conduct an in-service with the clinic's physical therapists and physical therapist assistants to ensure consistency with GFD education.
2. Therapists will be instructed to review the GFD documents with the participants.
3. The therapists will answer participant questions as appropriate.

During the course of the study: the INF® Therapy+ group will receive individual, face-to-face standardized verbal dietary education with weekly follow-up by a physical therapist either in person, via email, or over the phone. The INF® Therapy+ group will additionally receive meal preparation ideas and sample menus from the Gluten-Free Living website which promotes a gluten-free lifestyle. A co-investigator not involved in other participant assessments will complete these tasks] [For all participants] During the first visit, participants will be instructed verbally and in writing to report any unexpected medical care visits during the course of the study to the clinic via phone or email prior to any upcoming visits to allow for processing and re-scheduling. Therapists/student investigator will ask participants at the beginning of each session if they have had any unexpected visits to the urgent care, emergency department, physician, or surgeries. Should any adverse or serious adverse events (AE/SAE) be reported by the participants during enrollment in the study, the participant will not receive treatment or assessment that day, but be rescheduled.

* A NTC staff member (Jamie Hankins or Mark Bussell) will notify the student investigator (Criss Carlson) that same day if an AE or SAE occurs, and the principle investigator (Eric Johnson) will report the SAE/AE to the IRB in writing within the appropriate time limits established by the IRB.
* The principle investigator will notify the NTC in writing if the participant can continue with treatment or not within 24 to 48 hours.
* Participants may make up one missed session later in the same week or the following week after a missed session by receiving three INF® Therapy sessions within a week.
* If the patient returns and needs to be rescheduled for a second time, the patient will be dropped from the study.
* Should any participant miss treatment for more than seven consecutive days, they will be dropped from the study.

[All participants] Second assessment session for research purposes only (visit 12): Participants will return the week after completion of the ten INF® Therapy sessions for immediate post-intervention measurements. Participants will have opportunity to ask any questions they may have.

[Only for participants in the INF® Therapy+ group: For the INF® Therapy+ group, participants will be reminded to continue with dietary changes and follow up each week using the CDAT form. Participants will be contacted weekly by text message, e-mail, or phone call to facilitate compliance with the dietary changes. The evaluator (PT not involved in other participant assessments) will either assist participant in completing or review the CDAT questionnaire that the participant will be instructed to complete prior to the appointment each week. The weekly CDAT scores will be documented in a spreadsheet maintained separate from electronic medical records to keep principle evaluator blinded.

In order to accurately assess consistency, it may be ideal to randomly call or text massage participants by phone (with prior permission) each week with a reminder to complete the modified CDAT questionnaire.]

[All participants] Final assessment session for research purposes only (visit 13): At the end of three months post-INF® Therapy completion (10-14 weeks after second assessment), participants will return for post-intervention measurements. The post-intervention measurements will include Neuropad® neuropathy severity measure, MiniBESTest functional balance assessment, visual analog scale (VAS) for pain, the Celiac Dietary Adherence Test (CDAT), self-reported adherence to dietary changes questionnaire, the Pittsburg Sleep Quality Index (PSQI), International Physical Activity Questionnaire-short form (IPAQ-S), and State-Trait Anxiety Inventory Form Y (STAI-form Y).

After the three-month retesting, if a statistically significant difference emerges in the final analysis, then the INF® Therapy only group will be provided with the same dietary education materials the INF® Therapy+ group received.

ELIGIBILITY:
Inclusion Criteria

Participants in this study must be/have:

* Older adults between 50 to 75 years of age
* Willing to actively improve neuropathy symptoms
* Diagnosed with Type II diabetes
* Moderate to severe DPN (diabetic peripheral neuropathy) with symptoms below the knees of numbness, tingling, burning, sharp pain, and/or increased sensitivity
* Distal Symmetric Polyneuropathy (DSPN) form of DPN
* Independent in daily activities
* Do not use any assistive device for walking such as a cane, walker, or wheelchair

Exclusion Criteria

* Currently consuming a mainly plant-based or gluten-free diet
* Known allergy to chrome, nickel, or cobalt

Any of the following medical conditions:

* Current regimen of chemotherapy, radiation, or dialysis
* Lower extremity amputations and open wounds
* Documented active drug and/or alcohol misuse
* End stage renal failure
* End stage congestive heart failure
* Uncontrolled hypertension
* Chronic liver disease
* Advanced chronic obstructive pulmonary disease
* Active inflammations
* Other types of neuropathies not associated with diabetes including B12 deficiency
* Any other chronic medical conditions requiring active treatment
* Morbid obesity
* Pregnancy (self-reported)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Neuropathy Severity | Change between baseline and 3 Months post enrollment.
  The Neuropad® test measures sweat production as an indicator for peripheral neuropathy severity in people with type 2 diabetes. Sudometrics image analysis software will be utilized to analyze Neuropad® time to color change since it produces continuous outputs to quantify neuropathic severity.
Balance Stability | Change between baseline and 3 Months post enrollment.
  Mini balance evaluation system test (Mini-BESTest) assesses 4 balance-related subcategories of anticipatory, reactive postural control, sensory orientation, and dynamic gait, and takes approximately 15 minutes to administer.
Pain Intensity Level | Change between baseline and 3 Months post enrollment.
  The visual analog scale (VAS) for pain is a subjective measure of pain intensity.

SECONDARY OUTCOMES:
Gluten Consumption Assessment | Change between baseline and 3 Months post enrollment.
  The Celiac Dietary Adherence Test (CDAT) questionnaire gathers selected information on frequency of purposeful gluten consumption and self-efficacy to maintain compliance with a gluten-free diet.
Sleep Quality Assessment | Change between baseline and 3 Months post enrollment.
  The PSQI is a clinical questionnaire assessing quality of sleep and sleep disturbances over the past month. The questionnaire provides seven component scores assessing subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medications, and daytime dysfunction.
Total Weekly Physical Activity | Change between baseline and 3 Months post enrollment.
  The IPAQ-S measures intensity of physical activity and sitting time to estimate total physical activity per week.
State-Trait Anxiety Level | Change between baseline and 3 Months post enrollment.
  The STAI-form Y which is a definitive clinical measure of state and trait anxiety in adults.
Pain Quality Assessment | Change between baseline and 3 Months post enrollment.
  Pain Quality Assessment Scale (PQAS) is an adjusted version of the validated Neuropathic Pain Scale and includes 20 pain qualities and descriptors. The tool is validated for detecting changes in pre-post treatment pain quality and spatial characteristics of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Eric G Johnson, DSc, MS-HPEd, Principal Investigator — Department of Physical Therapy School of Allied Health Professions, Loma Linda University
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Worldwide toll of diabetes. Accessed January 20, 2020. https://www.diabetesatlas.org/en/sections/worldwide-toll-of-diabetes.html
- [Background] Cumulative confirmed COVID-19 deaths. Our World in Data. Accessed February 18, 2021. https://ourworldindata.org/grapher/cumulative-covid-deaths-region
- [Background] Feldman EL, Callaghan BC, Pop-Busui R, Zochodne DW, Wright DE, Bennett DL, Bril V, Russell JW, Viswanathan V. Diabetic neuropathy. Nat Rev Dis Primers. 2019 Jun 13;5(1):41. doi: 10.1038/s41572-019-0092-1. PMID 31197153
- [Background] Alshahrani A, Bussell M, Johnson E, Tsao B, Bahjri K. Effects of a Novel Therapeutic Intervention in Patients With Diabetic Peripheral Neuropathy. Arch Phys Med Rehabil. 2016 May;97(5):733-8. doi: 10.1016/j.apmr.2015.12.026. Epub 2016 Jan 22. PMID 26808781
- [Background] Bussell M. Neuropathic Treatment with Intraneural Facilitation. Presented at the: January 10, 2017. https://1drv.ms/p/s!AnT8e3KAvXUxgYc3Jf2Qkqu6HQb0lA?e=lHOOxP
- [Background] Role Of PT Diet Nutrition. APTA. Published September 20, 2019. Accessed November 13, 2020. https://www.apta.org/apta-and-you/leadership-and-governance/policies/role-of-pt-diet-nutrition
- [Background] Advocate | American Nutrition Association. Accessed November 13, 2020. https://theana.org/advocate
- [Background] Sahba K, Berk L, Bussell M, Lohman E, Zamora F, Gharibvand L. Treating peripheral neuropathy in individuals with type 2 diabetes mellitus with intraneural facilitation: a single blind randomized control trial. J Int Med Res. 2022 Aug;50(8):3000605221109390. doi: 10.1177/03000605221109390. PMID 35922961
- [Background] Zis P, Sarrigiannis PG, Rao DG, Hadjivassiliou M. Gluten neuropathy: prevalence of neuropathic pain and the role of gluten-free diet. J Neurol. 2018 Oct;265(10):2231-2236. doi: 10.1007/s00415-018-8978-5. Epub 2018 Jul 21. PMID 30032386
- [Background] Hadjivassiliou M, Sanders DS, Grunewald RA, Woodroofe N, Boscolo S, Aeschlimann D. Gluten sensitivity: from gut to brain. Lancet Neurol. 2010 Mar;9(3):318-30. doi: 10.1016/S1474-4422(09)70290-X. PMID 20170845
- [Background] Fleckenstein B, Qiao SW, Larsen MR, Jung G, Roepstorff P, Sollid LM. Molecular characterization of covalent complexes between tissue transglutaminase and gliadin peptides. J Biol Chem. 2004 Apr 23;279(17):17607-16. doi: 10.1074/jbc.M310198200. Epub 2004 Jan 27. PMID 14747475
- [Background] Jensen MP, Gammaitoni AR, Olaleye DO, Oleka N, Nalamachu SR, Galer BS. The pain quality assessment scale: assessment of pain quality in carpal tunnel syndrome. J Pain. 2006 Nov;7(11):823-32. doi: 10.1016/j.jpain.2006.04.003. PMID 17074624
- [Background] Galer BS, Jensen MP. Development and preliminary validation of a pain measure specific to neuropathic pain: the Neuropathic Pain Scale. Neurology. 1997 Feb;48(2):332-8. doi: 10.1212/wnl.48.2.332. PMID 9040716